CLINICAL TRIAL: NCT07327736
Title: Comparison Between Spontaneous Breathing-preserving Anesthesia and Double-lumen Endotracheal Intubation Anesthesia in Early-stage Non-small Cell Lung Cancer With a Diameter of ≤ 3 cm: a Prospective, Multicenter Randomized Controlled Study
Brief Title: Anesthesia Comparison in Early-stage Small NSCLC: A Multicenter RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT202508-17-KYB-15-XWK
Record Dates: First submitted 2025-12-11; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Patients With Suspected Non-small Cell Lung Cancer (NSCLC) at Clinical Stage T1
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Experimental): Non-intubated video-assisted thoracic surgery with spontaneous breathing (NIVATS)
  Interventions: Procedure: Non-intubated video-assisted thoracic surgery with spontaneous breathing (NIVATS)
- group B (Placebo Comparator): Tracheal Intubation with One-Lung Ventilation Group (OLV)
  Interventions: Procedure: Non-intubated video-assisted thoracic surgery with spontaneous breathing (NIVATS)

INTERVENTIONS:
Procedure: Non-intubated video-assisted thoracic surgery with spontaneous breathing (NIVATS) — NIVATS is a special method developed in the past two decades. It means that patients do not undergo tracheal intubation under general anesthesia during the entire surgical process, retaining their spontaneous breathing, but supraglottic airway devices (such as laryngeal masks, high-flow nasal catheters, mask ventilation) can be used to support their breathing. The purpose of this technology is to minimize the impact of general anesthesia, tracheal intubation, mechanical ventilation, etc. on patients.

SUMMARY:
This study is a prospective, randomized, controlled study, which intends to enroll patients with suspected early-stage NSCLC (non-small cell lung cancer) with a diameter of ≤ 3 cm as research subjects. The study is conducted in accordance with the Declaration of Helsinki. It has been approved by the Ethics Committee of the Second Affiliated Hospital of Air Force Medical University, and patients or their family members have signed the informed consent form. Patients undergoing VATS (video-assisted thoracic surgery) are enrolled in the Department of Thoracic Surgery of the Second Affiliated Hospital of Air Force Medical University. The patients are randomly divided into two groups: the NIVATS (non-intubated video-assisted thoracic surgery) group and the OLV (one-lung ventilation) group. By observing various perioperative indicators of the patients, the short-term efficacy of the two techniques in patients with early-stage NSCLC is compared, so as to evaluate the safety and effectiveness of the NIVATS surgical treatment method.

ELIGIBILITY:
Inclusion Criteria:

* Age ≤ 75 years;
* Gender is not limited;
* Patients with suspected T1 stage non-small cell lung cancer (NSCLC) in preoperative clinical staging, with thin-slice CT showing that the maximum tumor diameter is ≤ 3.0 cm, single or multiple nodules, and the nodules requiring surgical resection are located in the same ipsilateral lung lobe, with the number of nodules resected simultaneously ≤ 3;
* American Society of Anesthesiologists (ASA) classification ≤ Grade III (preferably Grade I - II is recommended);
* Eastern Cooperative Oncology Group (ECOG) performance status 0 - 1;
* Body Mass Index (BMI) < 25 kg·m-²;
* Normal cardiopulmonary function: predicted forced expiratory volume in the first second (FEV1%) > 50%, resting blood gas analysis showing arterial oxygen partial pressure (PaO2) ≥ 75 mmHg, arterial carbon dioxide partial pressure (PaCO2) < 45 mmHg; ejection fraction (EF) > 50%, 6-minute walk distance (6MWD) ≥ 350 m;
* No severe upper airway lesions, Mallampati classification I - II;
* No contraindications related to paravertebral nerve block and intercostal nerve block;
* Estimated surgical time ≤ 150 minutes;
* Patients have no history of clinically significant cardiac or neurological problems.

Exclusion Criteria:

* A history of ipsilateral lung surgery;
* Interstitial pneumonia, pulmonary fibrosis, severe emphysema, severe chronic obstructive pulmonary disease, acute phase of pulmonary infection, or uncontrolled asthma;
* Sleep apnea syndrome with anticipated airway difficulty or difficulty in airway management;
* Preoperative complications including coagulation dysfunction, hypoxemia, hypercapnia, or hepatic/renal insufficiency;
* Alteration of anesthesia or surgical plan;
* Persistent cough or increased risk of high airway secretion reflux;
* Mental disorders, inability to communicate, or refusal to sign the informed consent form;
* Participation in other clinical trials within 1 month before this trial;
* Those who are deemed unfit to participate in this trial by the researchers.

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 410 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Average postoperative hospital stay | up to 3 months
Intraoperative opioid consumption | 1 day

SECONDARY OUTCOMES:
Lung collapse score | 1 day
Intraoperative blood gas analysis (Q1h) | 1 day
Conversion to intubation rate | 1 day
Postoperative awakening time | 1 day
Time to first ambulation after surgery | up to 3 months
Ambulation rate within 4 hours after surgery | up to 3 months
Inflammatory markers (IL-6, peripheral neutrophil-to-lymphocyte ratio) | up to 3 months
Postoperative drainage volume | up to 3 months
Incidence of perioperative complications | up to 3 months
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0
15 item Quality of Recovery Rating Scale (QoR-15) | up to 1 year

OTHER OUTCOMES:
The impact of nursing education on discharge time and time to first ambulation after surgery | up to 3 months
Comparison of the effects of thoracic paravertebral nerve block and intrathoracic intercostal nerve block | up to 3 months
1-, 3-, and 5-year disease-free survival (DFS) | up to 5 years
1-, 3-, 5-, and 10-year overall survival (OS) | up to 10 years

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pompeo E, Mineo D, Rogliani P, Sabato AF, Mineo TC. Feasibility and results of awake thoracoscopic resection of solitary pulmonary nodules. Ann Thorac Surg. 2004 Nov;78(5):1761-8. doi: 10.1016/j.athoracsur.2004.05.083. PMID 15511470
- [Background] Pompeo E. State of the art and perspectives in non-intubated thoracic surgery. Ann Transl Med. 2014 Nov;2(11):106. doi: 10.3978/j.issn.2305-5839.2014.10.01. PMID 25489580
- [Background] Chiang XH, Lin MW. Converting to Intubation During Non-intubated Thoracic Surgery: Incidence, Indication, Technique, and Prevention. Front Surg. 2021 Oct 26;8:769850. doi: 10.3389/fsurg.2021.769850. eCollection 2021. PMID 34765639
- [Background] Lohser J, Slinger P. Lung Injury After One-Lung Ventilation: A Review of the Pathophysiologic Mechanisms Affecting the Ventilated and the Collapsed Lung. Anesth Analg. 2015 Aug;121(2):302-18. doi: 10.1213/ANE.0000000000000808. PMID 26197368
- [Background] Hung WT, Hung MH, Wang ML, Cheng YJ, Hsu HH, Chen JS. Nonintubated Thoracoscopic Surgery for Lung Tumor: Seven Years' Experience With 1,025 Patients. Ann Thorac Surg. 2019 Jun;107(6):1607-1612. doi: 10.1016/j.athoracsur.2019.01.013. Epub 2019 Feb 11. PMID 30763562
- [Background] Gelzinis TA, Sullivan EA. Non-Intubated General Anesthesia for Video-Assisted Thoracoscopic Surgery. J Cardiothorac Vasc Anesth. 2017 Apr;31(2):407-408. doi: 10.1053/j.jvca.2016.12.027. Epub 2016 Dec 23. No abstract available. PMID 28320572
- [Background] Janik M, Juhos P, Lucenic M, Tarabova K. Non-intubated Thoracoscopic Surgery-Pros and Cons. Front Surg. 2021 Dec 6;8:801718. doi: 10.3389/fsurg.2021.801718. eCollection 2021. PMID 34938770
- [Background] Liu J, Cui F, He J. Non-intubated video-assisted thoracoscopic surgery anatomical resections: a new perspective for treatment of lung cancer. Ann Transl Med. 2015 May;3(8):102. doi: 10.3978/j.issn.2305-5839.2015.04.18. PMID 26046043